CLINICAL TRIAL: NCT03814564
Title: ASSESSment of Peripheral Perfusion, Tissue Oxygen Saturation, Endothelial Function and Coagulation Disorder in Circulatory SHOCK, the ASSESS - SHOCK Study
Brief Title: ASSESSment of Perfusion, Oxygen Saturation, Endothelial Function and Coagulation in Circulatory SHOCK
Acronym: ASSESS-SHOCK
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Tampere University Hospital (Other); Kuopio University Hospital (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Erika Wilkman, MD PhD, Doctor, Adjunct Professor, Helsinki University Central Hospital
Other Study IDs: HUS/420/2018
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Circulatory Failure
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for later analysis of metabolomics, patient-related changes in biomarkers indicating endothelial and myocardial damage, coagulopathies and brain injury from consenting patients (such as syndecan-1 (SDC-1), vascular adhesion protein 1 (VAP1), CD73, heparin binding protein (HBP), endostatin, chromogranin, mitochondrial function tests and regulators (FGF-21 and GDF-15), blood count d-dimer, INR, neuron specific enolase). A separate sample for genetic analysis will be obtained that will be stored and processed further only if patient/next of kin provides the separately asked consent for the genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Circulatory failure / NIRS monitoring: Of the 400 patients, a subpopulation of the first 250 adult critically ill patients (≥18 years) requiring intensive care unit (ICU) care, including both surgical and medical ICU patients with circulatory shock will be included in the (near-infrared spectroscopy) NIRS-substudy.
  Interventions: Device: NIRS monitoring
- Circulatory Failure / no NIRS monitoring: Of the 400 patients, a subpopulation of the first 250 adult critically ill patients (≥18 years) requiring intensive care unit(ICU) care, including both surgical and medical ICU patients with circulatory shock will be included in the near-infrared spectroscopy (NIRS) substudy. All 400 patients will be analyzed for endotheliopathy incidence, metabolomics, genetic data (without NIRS monitoring). Representation of the study population will be ensured by enrolment of all consecutive patients at the study sites who meet the study enrollment criteria.
- Gut dysbiosis, delirium and long term cognition: ASSESS-shock participants that have been treated at Meilahti ICU:s and survived the ICU admission to discharge, who are living in the Helsinki and Uusimaa Hospital District area or reasonable traveling distance to the unit for cognitive testing.
  Cognitive function testing is performed after ICU discharge and at 3 and 6 months after ICU discharge. Testing of the microbiome is performed by collecting and analyzing fecal samples at ICU admission and at 7 days after ICU admission.

INTERVENTIONS:
Device: NIRS monitoring — Cerebral and peripheral NIRS monitoring of brain and tissue oxygenation. Of the 400 patients, a subpopulation of the first 250 adult critically ill patients (≥18 years) requiring ICU care, including both surgical and medical ICU patients with circulatory shock will be included in the NIRS-substudy. All 400 patients will be analyzed for endotheliopathy incidence, metabolomics, genetic data Representation of the study population will be ensured by enrolment of all consecutive patients at the study sites who meet the study enrollment criteria
  Groups: Circulatory failure / NIRS monitoring

SUMMARY:
The objective of the observational cohort study is (1) to deduce whether measurements of peripheral near-infrared spectroscopy (NIRS) (lower limb) associate with the development of organ dysfunction as assessed by daily Sequential Orfgan Failure Score (SOFA) in the Intensive Care Unit (ICU), (2)whether cerebral (frontal) tissue haemoglobin oxygen saturation (StO2) values are associated with delirium in the ICU and (3) the association of frontal and peripheral StO2 with other micro- and macrohemodynamic parameters in this patient group , (4) to deduce the associations between shock, endotheliopathy, disseminated intravascular coagulation (DIC) and tissue perfusion and, last, the feasibility of central and peripheral NIRS monitoring in shock patients in the ICU using the Medtronic INVOS NIRS StO2 appliances. In addition, the investigators target to evaluate (5) the incidence, evolution, and outcome of sepsis-associated DIC, and (6) the associations between a) continuous hemodynamic data, b) laboratory data (such as syndecan-1 (SDC-1), vascular adhesion protein 1 (VAP1), CD73, heparin binding protein (HBP), endostatin, chromogranin, mitochondrial function tests,blood count d-dimer, international normalized ratio (INR), neuron specific enolase and metabolomics data) (7) and study associations of singlenucleotide polymorphisms with developing organ dysfunction and 90-day mortality. To compare the hemodynamic alterations of burn patients to septic patients with the intention to find new ways to monitor and manage hemodynamic and particularly microcirculation in burn patients.

DETAILED DESCRIPTION:
Background:

Circulatory shock is a frequent condition in the intensive care unit, comprising roughly one of three patients in the intensive care unit (ICU), and associated with high mortality rates. Current treatment guidelines state that one of the main goals for therapeutic interventions is to improve tissue perfusion to prevent subsequent organ dysfunction and death. In acute critical illness, up to one fourth of the patients develop severe hemostatic aberrations and coagulopathy, called disseminated intravascular coagulation (DIC), which is associated with excess mortality.

Despite differences in the underlying cause, acutely critically ill patients share similar features that may be driven by shock. This response, potentially escalating to life-threatening conditions, is relatively homogenous. The shock induced sympatho-adrenal hyperactivation may be a critical driver this endotheliopathy. If allowed to proceed uncontrollably, damages to the microcirculation and organ dysfunction may follow.

Near-infrared spectroscopy (NIRS), a non-invasive method based on the principles of light transmission and absorption, offers a non-invasive and continuous bedside method to assess tissue haemoglobin oxygen saturation (StO2), which may serve as an indirect measure of the adequacy of tissue perfusion. NIRS could potentially be used for early identification of patients with tissue hypoperfusion and therefore high risk of developing organ dysfunction, and may also be used for assessing frontal cerebral oxygen saturation in circulatory failure and its use is well documented in general anaesthesia in many patient groups. There are some data showing an association between low frontal StO2 values and delirium in the ICU. The use of near-infrared spectroscopy to measure tissue oxygenation in healthy humans has been well validated. However, assessing tissue oxygenation using NIRS in critically ill patients is less well established. The hemodynamic and other systemic responses in burns are similar to those in septic shock. However, the mechanisms behind these responses have not been compared between burn and septic shock patients to our knowledge. Overall, the knowledge of microcirculation and how to monitor it in burn patients is limited.

Objectives:

The objective of the observational cohort study is (1) to deduce whether measurements of peripheral NIRS (lower limb registered proximal of the knee cap) associate with the development of organ dysfunction as assessed by daily sequential organ failure assessment score (SOFA) in the ICU during days 1 to 7 in the ICU, (2) whether cerebral (frontal) StO2 values are associated with delirium in the ICU and (3) the association of frontal and peripheral StO2 with other micro- and macrohemodynamic parameters in this patient group , (4) to deduce the associations between shock, endotheliopathy, DIC and tissue perfusion and, last, the feasibility of central and peripheral NIRS monitoring in shock patients in the ICU using the INVOS tm NIRS StO2 appliances. In addition, the investigators target to evaluate (5) the incidence, evolution, and outcome of sepsis-associated disseminated intravascular coagulation (DIC), and (6) the associations between a) continuous hemodynamic data, b) laboratory data (such as syndecan-1 (SDC-1), vascular adhesion protein 1 (VAP1), CD73, heparin binding protein (HBP), endostatin, chromogranin, mitochondrial function tests, blood count d-dimer, INR, neuron specific enolase and metabolomics data) (7) and study associations of singlenucleotide polymorphisms with developing organ dysfunction and 90-day mortality. To compare the hemodynamic alterations of burn patients to septic patients with the intention to find new ways to monitor and manage hemodynamic and particularly microcirculation in burn patients.

Design:

Observational multi-center study

Patient population:

Patients with circulatory shock admitted to the intensive care units (ICU) fulfilling the inclusion criteria.

Sample size:

A minimum of 250patients with circulatory shock with NIRS registration A minimum of 400 patients with sepsis for evaluation of incidence of DIC and metabolomics and genetic tests (genome-wide association study, GWAS)

Methods:

Patients with circulatory shock admitted to the intensive care unit (ICU) fulfilling the inclusion criteria but none of the exclusion criteria within 4 hours of vasopressor inititation in the ICU and signs of clinical hypoperfusion or elevated lactate levels. Frontal and peripheral NIRS StO2 registration is performed using the Medtronic INVOS appliances and bilateral central and peripheral sensors for 48 hours from study inclusion. The INVOS NIRS registration is blinded and cannot be used for clinical decision making. The frontal and peripheral StO2 registrations will be collected for further analyses. Blood samples will be taken from an arterial cannula at inclusion, and at 12 h, 24h and 48h, blood gas samples will be drawn every 2 hours. Data on demographic data, health status, chronic illnesses and medications prior to ICU admission will be collected during the study. Hemodynamic data, information on vasopressor and inotrope medication, need and use of sedatives, fluid balance and specific ICU interventions during the ICU stay will also be collected, as well as daily intensive care delirium screening checklist (ICDSC) and SOFA-score registrations. An electronic case report form (CRF) will be used in the study. In addition to clinical data, data of feasibility and reported problems considering the use of NIRS StO2 registrations will be collected. Blood samples will be frozen and stored locally for further processing and analyses.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 Critically ill patients requiring Intensive Care Unit (ICU) care with circulatory shock within 4 hours (≤ hours) of ICU admission or with circulatory shock developing in the ICU within 24 hours from ICU admission and within 4 hours of initiation of vasopressor treatment presenting with the below listed signs of for circulatory shock

1. Hypotension - need for vasopressor to achieve mean arterial pressure (MAP) ≥65 mmHg after 1L of crystalloid solution

   and
2. Any sign of hypoperfusion (at least one of the signs below)

   * blood lactate ≥2 mmol/L
   * mottling score ≥ 2
   * Base Excess (BE) ≤ - 5 mEq/L
   * prolonged capillary refill time ≥ 2 s
   * cool periphery beyond elbows or knees bilaterally
   * altered mentation

   OR

   Confirmed or suspected infection and anti-microbial treatment

   OR as an independent criteria for the ASSESS-SHOCK BURNS substudy
3. Burn injury ≥30% total body surface area(TBSA), ICU admission within 12h of the injury, with or without hypotension and signs of hypoperfusion within 4 hours of ICU admission

Exclusion Criteria:

* Age < 18 years
* Pregnant or lactating
* Known refusal to any clinical study or this specific study
* Consent not obtained (according to local regulatory statements for ethical conduct of research)
* Out-of-hospital cardiac arrest (OHCA) patients
* Terminal illness and not considered for full intensive care support
* Planned postoperative admission
* Postoperative intensive care after organ transplantation
* Patients who are likely to be transferred to the ward in 24 hours
* Defects of skin, underlying tissues or extremities preventing the use of the central or peripheral NIRS probes (the first 250 enrolled patients)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise 400 critically ill patients with circulatory shock from 4 university hospitals during approximately 2 years between April 2019 and December 2021. Of the 400 patients, a subpopulation of the first 250 adult critically ill patients (≥18 years) requiring ICU care, including both surgical and medical ICU patients with circulatory shock will be included in the NIRS-substudy. All 400 patients will be analyzed for endotheliopathy incidence, metabolomics, genetic data (without NIRS monitoring). Representation of the study population will be ensured by enrolment of all consecutive patients at the study sites who meet the study enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in severity of Organ dysfunction during the first week in ICU (study period) | At 7 days in ICU
  Change in the total Sequential Organ Failure Assessment (SOFA) score from day 1 to day 7 in the ICU, higher SOFA score indicates greater severity of organ failure, the total SOFA score ranges from 0-24 points
Average severity of Organ dysfunction during the first 7 days in the ICU (study period) | First week in the Intensive Care Unit after admission
  Average Sequential Organ Failure Assessment (SOFA) during days 1 to day 7 in the ICU, higher SOFA score indicates greater severity of organ failure, the total SOFA score ranges from 0-24 points
New organ dysfunctions | First week in the Intensive Care Unit after admission
  Number of new organ dysfunctions (new organ dysfunction defined as one of 6 SOFA subscores ≥3 points/ total 4 points, higher points indicate greater severity. Only one new organ dysfunction / each subscore can be used for calculation of total number of new organ dysfunctions in one week
90-day mortality | 90 days
  Death within 90 days from ICU admission

SECONDARY OUTCOMES:
Intensive care delirium incidence | First week in the Intensive Care Unit after admission
  Delirium diagnosis in the ICU assessed by Intensive Care Delirium Scoring Checklist (ICDSC) scoring during days 1-7 defined as ICDSC score value of four points or more ( total score: 0-8 points)
Intensive care delirium severity | First week in the Intensive Care Unit after admission
  Number of Intensive Care Delirium Scoring Checklist (ICDSC) scores (assessment performed twice daily) of ≥4 points indicating presence of delirium during days 1-7
Intensive care delirium scoring checklist aggregate and average score during first week in intensive care | First week in the Intensive Care Unit after admission
  Aggregate Intensive Care Delirium Scoring Checklist (ICDSC) scores during days 1-7 . Total score ranges from 0 to 8 points. The aggregate score of all daily ICDSC measurements ( sum of all daily scores performed twice daily) will be divided by number of measurements to adjust for possible differences in number of measurements (= average ICDSC score)
INVOS NIRS feasibility and safety questionnaire | 0-48 hours in Intensive Care Unit after enrolment into study
  Feasibility of frontal and peripheral near-infrared spectroscopy tissue (NIRS) haemoglobin oxygen saturation (StO2) assessment in circulatory shock during the 48 h registration. Feasibility and registration issues are assessed using a questionnaire. Feasibility will be assessed every eight hours ( during each nurse's shift assessing feasibility and saefty on a scale from 0 to 5. Higher score indicatesmore severe feasibility issues
Time to Extubation | 28 days
  Time to extubation
Days off ventilator in 28 days | 28 days
  Days off ventilator in 28 days
Days without vasoactive medication in 28 days | 28 days
  Days without vasopressor or inotropic medication
Days without RRT in 28 days | 28 days
  Days without renal replacement therapy of any kind in 28 days
ICU length of stay | 90 days
  ICU length of stay
28-day mortality | 28 days
  28-day mortality
Cognitive dysfunction after ICU discharge | 6 months
  Cognitive dysfunction assessed by a set of neuropsychological tests

OTHER OUTCOMES:
Glycocalyx and endothelial injury biomarkers such as: Syndecan-1 (SDC-1), vascular adhesion protein 1 (VAP1), CD73, heparin binding protein (HBP), angiopoietin-2, endostatin, chromogranin | First week in the Intensive Care Unit after admission
  Injury of the endothelium and glycocalyx

CONTACTS AND LOCATIONS:
Overall Officials: Erika Wilkman, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varis E, Heliste M, Hastbacka J, Vaara ST, Skrifvars MB, Pettila V, Laaperi M, Kuitunen A, Vahtera A, Wilkman E. Clinical outcomes and peripheral tissue oxygen saturation monitoring of the knee region by near-infrared spectroscopy in circulatory shock: a prospective observational cohort study. Crit Care. 2025 Mar 19;29(1):125. doi: 10.1186/s13054-025-05363-1. PMID 40108719